CLINICAL TRIAL: NCT06439225
Title: A Randomized Phase III Trial Investigating Platinum and Taxane Chemotherapy in Metastatic Castration Resistant Prostate Cancer Patients With Alterations in DNA Damage Response Genes
Brief Title: Platinum and Taxane Chemo in Met Castration Resistant Prostate Cancer Patients With Alterations in DNA Damage Response Genes
Acronym: OPTION-DDR
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR25
Record Dates: First submitted 2024-05-27; First posted 2024-06-03 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Castration-resistant Prostate Cancer; Metastatic Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Docetaxel (Active Comparator)
  Interventions: Drug: Docetaxel
- Carboplatin + Docetaxel (Experimental)
  Interventions: Drug: Docetaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Docetaxel — 75mg/m2 q21 days
Drug: Carboplatin — AUC5 q21 days
  Arms: Carboplatin + Docetaxel

SUMMARY:
The usual approach for most patients who are not in a study is treatment with docetaxel.

This study is being done to answer the following question: Can the chance of prostate cancer growing or spreading be lowered by adding a drug to the usual approach?

This study is being done to find out if this approach is better or worse than the usual approach for prostate cancer. The usual approach is defined as the care most people get for prostate cancer.

DETAILED DESCRIPTION:
If taking part in this study, the patient will either get docetaxel, or carboplatin in addition to docetaxel. In both cases, the cancer will be monitored by CT scans and bone scans every 9 weeks, and blood tests every 3 weeks. Study treatments, scans, and tests will continue until the disease gets worse.

After finishing study treatment, even if treatment is stopped before the disease gets worse, the study doctor will continue to follow patients condition, watch for side effects and keep track of the health of the patient. If treatment is stopped before the disease got worse, patients will be asked to continue getting CT scans and bone scans every 9 weeks, and blood tests every 3 weeks, until the disease worsens. If the disease gets worse while receiving treatment, or after treatment is stopped, the patient will be contacted by phone every 3 months for the rest of their life to monitor their status. Patients may be seen more often if the study doctor thinks it is necessary.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of adenocarcinoma of the prostate. The presence of neuroendocrine or small cell carcinoma will be exclusionary
* Prior treatment with any ARPI, such as abiraterone, enzalutamide, apalutamide, or darotlutamide, is required.
* Participants must have recovered to ≤ grade 1 from all reversible toxicity related to prior systemic or radiation therapy, with the exception of chemotherapy induced alopecia and grade 2 peripheral neuropathy, and have adequate washout as follows:
* Longest of one of the following:

  * Two weeks or 5 half lives (whichever is longer) for oral therapies (such as abiraterone, apalutamide, enzalutamide, darolutamide and olaparib)
  * Standard cycle of standard IV or IM therapies (such as radium 223 or Lu-177-PSMA-617
  * 2 weeks, 5 half lives, or standard cycle length (whichever is longer) for investigational agents
* Previous major surgery is permitted provided that surgery occurred at least 28 days prior to participant enrollment and that wound healing has occurred
* Prior external beam radiation is permitted provided a minimum of 7 days have elapsed between the last dose of radiation and date of enrollment
* Radiologically documented presence of metastatic disease within 28 days prior to randomization
* Disease progression after ARPI therapy as assessed by the investigator with at least one of the following:
* PSA progression with a minimum of two rising PSA values at least 1 week apart, at least 25% and 2ug/L above baseline/nadir.
* Radiographic progression of soft tissue disease by RECIST 1.1 criteria or bone metastases by PCWG3 criteria.
* Medical or surgical castration with serum testosterone levels <50ng/dL or <1.7mmol/L
* Qualifying Tier I or Tier II (clinically significant/likely clinically significant or pathogenic / likely pathogenic) germline or somatic alterations involving one or more of the following DDR genes: BRCA1, BRCA2, ATM, ATR, BRIP1, BARD1, CDK12, CHEK1, CHEK2, ERCC2, FANCA, FANCC, FANCD2, FANCL, PALB2, RAD51B, RAD51C, RAD51D, RAD54L. Monoallelic gene deletions in isolation will not be eligible.
* Age 18 years or older.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 2
* Participants must have adequate organ and marrow function measured within 14 days prior to enrolment
* Life expectancy > 12 weeks.
* If the participant and the participant's partner are of childbearing potential, they must agree to use medically accepted methods of contraception (e.g., barrier methods, including male condom, female condom, or diaphragm with spermicidal gel) during the course of the study and for 6 months after the last dose of study drug.
* Participant is able (i.e. sufficiently fluent) and willing to complete the quality of life and health utility questionnaires in either English or French
* Participant consent must be appropriately obtained in accordance with applicable local and regulatory requirements. Each participant must sign a consent form prior to enrollment in the trial to document their willingness to participate.
* Participants must be accessible for treatment and follow-up. Investigators must assure themselves the participants enrolled on this trial will be available for complete documentation of the treatment, adverse events, and follow-up.
* In accordance with CCTG policy, protocol treatment is to begin within 2 working days after participant enrolment.

Exclusion Criteria:

* Received prior platinum chemotherapy (i.e. carboplatin, cisplatin, oxaliplatin, satraplatin) at any time; received prior taxane chemotherapy (docetaxel, paclitaxel, cabazitaxel) with the exception of docetaxel for mCSPC as long as it was no more than 6 cycles and at least 12 months have elapsed from their last treatment to the date of enrollment.
* Active anticancer systemic therapy or investigational agents within 14 days of randomization.
* Uncontrolled intercurrent illness including, but not limited to: active infection, symptomatic congestive heart failure (NYHA Class III or IV heart disease), unstable angina pectoris, cardiac arrhythmia, uncontrolled hypertension or psychiatric illness/social situations that would limit compliance with study requirements.
* Participants with myelodysplastic syndrome/acute myeloid leukemia.
* Malignancy within the previous 2-years with a > 30% probability of recurrence within 12 months, with the exception of non-melanoma skin cancer, and in-situ or superficial bladder cancer.
* Participants with known symptomatic brain metastasis. However, participants with asymptomatic, treated brain metastases that have been stable for at least 12 weeks are eligible for study entry.
* Participants with symptomatic or impending cord compression unless appropriately treated beforehand and clinically stable and asymptomatic.
* Presence of a condition or situation, which, in the investigator's opinion, may put the participant at significant risk, may confound the study results, or may interfere significantly with participation in the study.
* Live attenuated vaccination administered within 30 days prior to randomization.
* For participants with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated. Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. For participants with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* Unable to obtain provincial reimbursement of carboplatin and docetaxel

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 236 (Estimated)
Dates: Start 2024-12-30 (Actual); Primary Completion 2029-09-30 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 5.25 years

SECONDARY OUTCOMES:
To compare the two treatment arms with respect to PSA response | 5.25 years
  Defined as a reduction in PSA from baseline by 50%
To compare the two treatment arms with respect to progression free survival | 5.25 years
  as defined by PCWG3 and RECIST 1.1
To compare the two treatment arms with respect to time to next systemic therapy | 5.25 years
To compare the two treatment arms with respect to time to number and severity of adverse events | 5.25 years
  Utilizing CTCAE version 5.0
To compare the two treatment arms with respect to patient-reported Quality of Life (QoL) quantified by FACT-P questionnaire | 5.25 years
To compare the two treatment arms with respect to patient-reported Quality of Life (QoL) quantified by FACT-Taxane questionnaire | 5.25 years
To compare the two treatment arms with respect to patient-reported Quality of Life (QoL) quantified by BPI-SF questionnaire | 5.25 years
Economic Evaluation of healthcare utilization | 5.25 years
  Health system resources will be identified as, but not limited to, clinic visits, treatments (radiation, surgery, medication), physician encounters, hospitalizations related to treatment and complications, emergent visits and diagnostics.
Economic Evaluation of health utilities measured by Eq-5D-5L | 5.25 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kolinsky, Study Chair — Cross Cancer Institute, Edmonton, Alberta, Canada
Locations (14):
- Canada (14):
  - Arthur J.E. Child Comprehensive Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA - Vancouver, Vancouver, British Columbia
  - William Osler Health System, Brampton, Ontario
  - Waterloo Regional Health Network (WRHN), Kitchener, Ontario
  - London Health Sciences Centre Research Inc., London, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Odette Cancer Centre, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - CHUM-Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - The Jewish General Hospital, Montreal, Quebec
  - CHU de Quebec-Hopital l'Enfant-Jesus (HEJ), Québec, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: Yes
As per CCTG policy
URL: https://www.ctg.queensu.ca/docs/public/policies/DataSharingandAccessPolicy.pdf